CLINICAL TRIAL: NCT03077516
Title: Post-Market, Long-Term Follow Up of Mobi-C® Cervical Disc for One and Two Level Treatment of Cervical Disc Disease
Status: Completed | Type: Observational
Sponsor: LDR Spine USA (Industry)
Responsible Party: Sponsor
Other Study IDs: MC-100
Record Dates: First submitted 2016-11-28; First posted 2017-03-13 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Cervical Disc Disease; Cervical Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Mobi-C: Prior recipient of Mobi-C Disc in IDE/Post Approval Study
  Interventions: Device: Mobi-C
- ACDF: Prior control subject in IDE/Post Approval Study

INTERVENTIONS:
Device: Mobi-C — Device for cervical intervertebral disc replacement at one or two contiguous levels
  Other Names: Mobi-C Cervical Disc Prosthesis
  Groups: Mobi-C

SUMMARY:
The purpose of this study is to evaluate clinical and patient-reported outcomes at 10 years following surgery for a cohort of Mobi-C subjects treated on the IDE/Post Approval studies

DETAILED DESCRIPTION:
This is a prospective, multi-center, consecutive cohort study. Subjects invited to participate in this study will have completed the Mobi-C IDE study (G050212). In this study, five hundred and seventy-five subjects were randomized to either the Mobi-C prosthesis or the control treatment - conventional anterior cervical discectomy and fusion (ACDF) with anterior cervical plating. The study was randomized in a 2 to 1 ratio (two Mobi-C subjects for every one subject receiving ACDF with anterior cervical plate). The subject retention rate for Mobi-C subjects was 80.1% (1 level)-84.4% (2 level) at 7 years.

As non-inferiority (1-level) and superiority (2-level) have been well established through 7 years, the design of this study will focus on the long-term outcomes of a cohort of the Mobi-C arm of the study and evaluate the durability of outcomes at 10 years. Study sites invited to participate will be those that enrolled at least 10 subjects, and also had the highest retention rates at 7 years (≥70%). All subjects at these sites will be contacted to participate in an additional 10 year follow up visit. It is estimated that up to 250 subjects will be enrolled at 9-12 study sites.

Certain endpoints are better assessed in comparison to the control ACDF arm, such as adjacent segment degeneration and subsequent surgery. This study has been amended to include a subset of sites that will also enroll control subjects. Up to 3 sites and 50 subjects will be included in this control cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Prior enrollment in LDR-001 Pivotal Study (IDE G050212);
2. Written informed consent provided by subject or subject's legally authorized representative

Exclusion Criteria:

1. Documented withdrawal of consent from prior Mobi-C study;
2. Documented non-compliance (including unwillingness to return to the site for follow-up visits)
3. Reported pregnancy at time of enrollment, or with plans to become pregnant prior to completing study X-Rays

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mobi-C and control subjects treated on the IDE/Post Approval studies, with one or two level disc replacement
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
NDI Score | 10 Years

SECONDARY OUTCOMES:
Overall Success | 10 Year
  Composite score composed of: 1) NDI improvement of at least 15 points (out of 50) from baseline; 2) No subsequent surgical intervention at the index level or levels; 3) No potentially (possibly or probably) device-related adverse event; 4) Maintenance or improvement in all components of neurologic status; and 5) No Mobi-C intraoperative changes in treatment.
Neck Pain/Arm Pain VAS | 10 Year
QOL SF-12 | 10 Year
Patient Satisfaction | 10 Year
  Measured by a two questions scale that includes ranking of level of satisfaction and willingness to recommend treatment.
Secondary surgery Rate | 10 Years
Device related complications | 10 Years
Device displacement or migration | 10 Year
  Radiographic assessment of movement of device from original placement
Range of motion | 10 Years
  Radiographically measured angle, in degrees, between endplates of adjacent vertebrae
Disc Height | 10 Years
  Radiographically measured distance, in mm, from corner of superior vertebra to corresponding corner of inferior vertebra
Heterotopic Ossification | 10 Years
  Qualitative radiographic assessment using McAfee grading system, grades 1-4
Adjacent Segment Degeneration | 10 Years
  Qualitative radiographic assessment using Kellgren-Lawrence Disc Degeneration Grading, grades 0-IV

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Orange County Neurosurgical Associates, Laguna Hills, California
  - Desert Orthopedic Center, Rancho Mirage, California
  - UC Davis Spine Center, Sacramento, California
  - The Spine Institute, Santa Monica, California
  - Orthopedics Northeast, Fort Wayne, Indiana
  - Spine Institute of Louisiana, Shreveport, Louisiana
  - Texas Back Institute, Plano, Texas
  - Texas Spine and Joint Hospital, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Radcliff K, Coric D, Albert T. Five-year clinical results of cervical total disc replacement compared with anterior discectomy and fusion for treatment of 2-level symptomatic degenerative disc disease: a prospective, randomized, controlled, multicenter investigational device exemption clinical trial. J Neurosurg Spine. 2016 Aug;25(2):213-24. doi: 10.3171/2015.12.SPINE15824. Epub 2016 Mar 25. PMID 27015130
- [Background] Hisey MS, Zigler JE, Jackson R, Nunley PD, Bae HW, Kim KD, Ohnmeiss DD. Prospective, Randomized Comparison of One-level Mobi-C Cervical Total Disc Replacement vs. Anterior Cervical Discectomy and Fusion: Results at 5-year Follow-up. Int J Spine Surg. 2016 Feb 26;10:10. doi: 10.14444/3010. eCollection 2016. PMID 27162712
- [Background] Jackson RJ, Davis RJ, Hoffman GA, Bae HW, Hisey MS, Kim KD, Gaede SE, Nunley PD. Subsequent surgery rates after cervical total disc replacement using a Mobi-C Cervical Disc Prosthesis versus anterior cervical discectomy and fusion: a prospective randomized clinical trial with 5-year follow-up. J Neurosurg Spine. 2016 May;24(5):734-45. doi: 10.3171/2015.8.SPINE15219. Epub 2016 Jan 22. PMID 26799118
- [Background] Ament JD, Yang Z, Nunley P, Stone MB, Lee D, Kim KD. Cost Utility Analysis of the Cervical Artificial Disc vs Fusion for the Treatment of 2-Level Symptomatic Degenerative Disc Disease: 5-Year Follow-up. Neurosurgery. 2016 Jul;79(1):135-45. doi: 10.1227/NEU.0000000000001208. PMID 26855020